CLINICAL TRIAL: NCT06787885
Title: Evaluation of Efficacy and Safety Parameters of Different Antibiotics Regimens for Management of Empyema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Mohamed, Teaching assistant, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M721
Record Dates: First submitted 2025-01-13; First posted 2025-01-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Empyema, Pleural
MeSH Terms: conditions — Empyema, Pleural | interventions — Levofloxacin; Clindamycin; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patient with empyema (Other): Tavanic (levofloxacin )and dalacin (clindamycin)
  Interventions: Drug: Levofloxacin + cefipime
- Empyema patient (Other): Tavanic (levofloxacin) and cefipime
  Interventions: Drug: Levofloxacin + clindamycin
- patient has lung empyema (Other): Moxiflox (moxifloxacin) and meronem
  Interventions: Drug: Moxifloxacin + meronam

INTERVENTIONS:
Drug: Levofloxacin + clindamycin — Group 1
  Arms: Empyema patient
Drug: Levofloxacin + cefipime — Group 2
  Arms: Patient with empyema
Drug: Moxifloxacin + meronam — Group 3
  Arms: patient has lung empyema

SUMMARY:
To evaluate the impact of using different antibiotic regimens including single and combined agents as the empirical therapy and evaluate the clinical outcomes regarding safety, efficacy, and pharmacodynamics parameters.

ELIGIBILITY:
Inclusion Criteria:

Confirmed Diagnosis of Empyema: Patients with a clinical and radiological diagnosis of

Exclusion Criteria:

1 - Hypersensitivity or Allergy to the selected antibiotic: Patients with a known history of hypersensitivity or allergic reactions to used antibiotics.

2- Pregnancy and Lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Evalutate different antibiotics | 2 weeks
  To evaluate the impact of using different antibiotic regimens including single and combined agents as the empirical therapy .

CONTACTS AND LOCATIONS:
Overall Officials: Raghda Roshdy Hussein, Assistant professor, Study Chair — Faculty of pharmacy Beni suef University; Marwa Kamal Tolba, Assistant professor, Study Director — Faculty of pharmacy Fayoum University; Yassmin Mohamed Medany, Lecturer, Study Director — Faculty of pharmacy Benisuef University; Mona Ibrahim Ahmed, Assistant professor, Study Director — Faculty of Medicine Fayoum University; Abdelrahman Ahmed Mohamed, Teaching assistant, Principal Investigator — Faculty of pharmacy Fayoum University
Locations (1):
- Fayoum University hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided